CLINICAL TRIAL: NCT00989885
Title: The Effectiveness of the Epworth´s Sleepiness Scale as a Resource Aid in the Diagnosis of the Syndrome of Obstructive Sleep Apnea
Brief Title: ESS as a Diagnosis Resource Aid of the Syndrome of Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Collaborators: CESF - Centro de Estudos do Sono de Fortaleza LTDA (Unknown)
Responsible Party: Ingrid Correia Nogueira, Fortaleza University
Other Study IDs: FR132544
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Sleep Apnea; Mixed Central and Obstructive Sleep Apnea; Sleep-Disordered Breathing
Keywords: Evaluation; Obstructive sleep apnea; Polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obstructive Sleep Apnea: 475 patients that sought the CESF to probable diagnosis of some sleep disorder, subsequently diagnosed with Obstructive Sleep Apnea.
  Interventions: Other: Questionnaire and polysomnography

INTERVENTIONS:
Other: Questionnaire and polysomnography — Comparison of polysomnography data records and previously made questionnaire, with the Epworth Sleepiness Scale.

SUMMARY:
The aim of this study was to analyze the effectiveness of the Epworth's sleepiness scale as a recourse aid in the diagnosis of the syndrome of obstructive sleep apnea. 475 patients attended this study, that sought the CESF to probable diagnosis of some sleep disorder. The data were collected from records, wich are of questionnaires, including the ESE, prepared by the CESF professionals and responded, previously, by the own patients. The study compared the result obtained in the scale of Epworth with the data of polysomnography. The analysis of data was performed using the SPSS, based on descriptive and inferential statistics, being used the average considering the standard deviation, and, to the crossing of variables, was used the chi-square test of Pearson, considering as significant statistically values of p<0.05. The results showed that gender, age and BMI are predisposing factors to SOSA.

ELIGIBILITY:
Inclusion Criteria:

* Charts of whose admission of patients was from October 2005 to July 2007
* Patients referred to the CESF for possible diagnosis of a sleep disorder

Exclusion Criteria:

* incomplete data
* patients with concomitant diseases (heart disease, hormonal disease, chronic obstructive pulmonary disease and neurological patients)
* patients undergoing uvulopalatopharyngoplasty

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that sought the CESF to probable diagnosis of some sleep disorder
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Epworth's sleepiness scale | March 2007

SECONDARY OUTCOMES:
Polysomnography | May 2007

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid C Nogueira, Bachelor, Principal Investigator — Fortaleza University; Ana Cristhina O Brasil, Master, Study Director — Fortaleza University; Priscilla O Azevedo, Bachelor, Principal Investigator — Fortaleza University; Vera Maria A Lacerda, Bachelor, Principal Investigator — Fortaleza University
Locations (1):
- Fortaleza University - Nucleus of Integrated Medical Attention, Fortaleza, Ceará, Brazil